CLINICAL TRIAL: NCT06212804
Title: A Phase 1, Randomized, Placebo-controlled, Double Blind, Single Ascending Dose, First-in-human Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of VIS954 in Healthy Male and Female Participants
Brief Title: A Study to Investigate the Safety, Pharmacokinetics, and Pharmacodynamics of VIS954 in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Visterra, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VIS954-101
Record Dates: First submitted 2023-12-11; First posted 2024-01-19 (Actual); Results first posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-06

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Intervention Model Description: Phase 1, randomized, placebo-controlled, double-blind, single ascending dose study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- VIS954 Dose 1 (Experimental): A single VIS954 Dose 1 will be administered subcutaneously on Day 1
  Interventions: Biological: VIS954
- VIS954 Dose 2 (Experimental): A single VIS954 Dose 2 will be administered subcutaneously on Day 1
  Interventions: Biological: VIS954
- VIS954 Dose 3 (Experimental): A single VIS954 Dose 3 will be administered subcutaneously on Day 1
  Interventions: Biological: VIS954
- VIS954 Dose 4 (Experimental): A single VIS954 Dose 4 will be administered subcutaneously on Day 1
  Interventions: Biological: VIS954
- VIS954 Dose 5 (Experimental): A single VIS954 Dose 5 will be administered subcutaneously on Day 1
  Interventions: Biological: VIS954
- VIS954 Dose 6 (Experimental): A single VIS954 Dose 6 will be administered subcutaneously on Day 1
  Interventions: Biological: VIS954
- Placebo (Placebo Comparator): A single Placebo dose will be administered subcutaneously on Day 1 for 2 participants in each cohort.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: VIS954 — A humanized IgG4 monoclonal antibody.
  Arms: VIS954 Dose 1; VIS954 Dose 2; VIS954 Dose 3; VIS954 Dose 4; VIS954 Dose 5; VIS954 Dose 6
Other: Placebo — VIS954 Placebo
  Arms: Placebo

SUMMARY:
This is a first-in-human (FIH), randomized, placebo-controlled, double-blind, single ascending dose (SAD) study to assess the safety and tolerability of VIS954, a monoclonal antibody, in healthy adult male and female participants.

DETAILED DESCRIPTION:
The study will be conducted in 6 sequential cohorts. Each cohort will enroll 9 participants, randomized to VIS954 or placebo at a ratio of 7:2.

On Day 1, a single dose of VIS954 or placebo will be administered SC. Sentinel participants will be utilized in each cohort. After 14 days, the safety data will be evaluated and a decision to admit and dose the next cohort will be made.

The total duration of the clinical study per participant will be up to 102 days (approximately 4 months).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participant between 18 to 55 years of age, inclusive, at the screening visit.
2. Non-Japanese participant: Participant does not meet the criteria specified below for 'Japanese Participant'.
3. Japanese participant: Participant is of Japanese descent as evidenced by verbal confirmation of familial heritage (a participant's 4 grandparents were born in Japan and recognized to be 'Japanese').
4. Body mass index between 18.0 and 30.0 kg/m2, inclusive, at the screening visit.
5. Total body weight between 50.0 and 120.0 kg, inclusive, at the screening visit.
6. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and the protocol.
7. Willing and able to participate in the study for the defined duration of the study.
8. Female participants will be nonpregnant, nonlactating, and either postmenopausal for at least 1 year or surgically sterile for at least 3 months, or will agree to use highly effective methods of contraception from the period prior to study enrollment until 30 days after Day 56; women of childbearing potential must have a negative serum beta-human chorionic gonadotropin (β-hCG) test at screening and a negative urine pregnancy test at baseline prior to administration of the study intervention.
9. Male participants with female partners of childbearing potential must agree to use double barrier contraception or abstain from sex during the study and until 90 days after Day 56. Male participants must agree to refrain from sperm donation for the duration of the study and until 90 days after Day 56. This criterion may be waived for male participants who have had a vasectomy greater than 6 months prior to enrollment.
10. Healthy, as determined by prestudy medical evaluation (medical history, physical examination, vital signs, 12-lead ECG, and clinical laboratory evaluations), as judged by the principal investigator.

Exclusion Criteria:

1. Participant has a history or current evidence of a serious and/or unstable cardiovascular, respiratory, gastrointestinal, hematologic, autoimmune, blood dyscrasias or other medical disorder, including psychiatric disorders, cirrhosis, or malignancy. History of minor skin cancers (not including melanoma) or surgically treated, limited cervical carcinomas (ie, carcinoma in situ) are not exclusionary.
2. Participant is participating in another clinical study of any investigational drug, device, or intervention or has received any investigational medication during the last 30 days or 5 half-lives, whichever is longer, before baseline (Day -1).
3. Previous receipt of antibody or biologic therapy.
4. History of a previous hypersensitivity or severe allergic reaction with generalized urticaria, angioedema, or anaphylaxis to any of the ingredients of the VIS954 SC injection formulation.
5. Blood pressure > 160/100 mmHg or < 90/50 mmHg (may be repeated once if abnormal), at the screening visit or Day -1.
6. History of any infection requiring hospitalization or treatment with antivirals, antibiotics, or systemic antifungals within 3 months prior to screening.
7. Received a vaccination, other than COVID-19 vaccination, during the 30 days prior to administration of the first dose of study intervention. A COVID-19 vaccination cannot be received within 7 days prior to the first dose of study intervention and until 14 days after the last dose.
8. Has received any prescription or nonprescription (over-the-counter) medication during the last 30 days or 5 half-lives, whichever is longer, preceding baseline (Day -1), with the exception of acetaminophen, ibuprofen, naproxen (or other over-the-counter nonsteroidal anti-inflammatory drugs [NSAID]), hormonal contraceptives, topical medications, vitamins, and dietary or herbal remedies.
9. Any participant who has a recent history of alcohol or drug/chemical abuse, at the discretion of the investigator, will be excluded.
10. Enrolled participants must abstain from consumption of nicotine containing products from Day -1 through discharge.
11. Enrolled participants must abstain from consumption of cannabinoids from Day-1 through end of study.
12. For the duration of the study, enrolled male participants should not consume more than 15 standard drinks per week (7 days) and female participants should not consume more than 10 standard drinks per week (7 days). A standard drink equals 10 g of alcohol. Enrolled participants must abstain from consuming alcohol 48 hours prior to check-in on Day -1 through discharge.
13. Participant with a positive urine drug or alcohol breath screen test result at screening or Day -1. The urine drug screen and alcohol breath screen may be repeated once at the discretion of the investigator. The urine drug screen also screens for methylenedioxymethamphetamine and propoxyphene. If a participant tests positive on these tests, inclusion of that participant into the study will be based on the principal investigator's judgment with consultation, as needed, with the medical monitor and the sponsor.
14. Any chronic infectious disease (eg, chronic urinary tract infection, chronic sinusitis, bronchiectasis, active pulmonary or systemic tuberculosis [TB], chronic viral hepatitis such as hepatitis C or hepatitis B, or human immunodeficiency virus [HIV] infection).
15. Participant who has donated > 500 mL of blood within 60 days prior to start of the screening visit or the participant has donated any plasma within 7 days prior to baseline (Day -1).
16. Coronavirus disease 2019:

    * Current symptoms of infection.
    * Diagnosis of COVID-19 (reverse transcription polymerase chain reaction [RT-PCR], antigen testing, or clinical diagnosis) in the 21 days prior to screening.
    * Ongoing diagnosis of "Long-COVID" symptoms, due to a prior COVID-19 infection.
17. Is an employee of the clinical research team (any sponsor or research site employee), or has a family member who is an employee of these organizations.
18. Participant is judged by the investigator or the medical monitor to be inappropriate for the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2023-11-21 (Actual); Primary Completion 2024-07-19 (Actual); Study Completion 2024-07-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Visterra Clinical Site, Anaheim, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase 1, double-blind, single ascending dose, first-in-human study was conducted in healthy participants at a single investigational site.
Pre-assignment Details: The study was conducted in 6 sequential cohorts. In each cohort, participants were randomized in a 7:2 ratio to receive VIS954 or matching placebo. The study consisted of a screening period (up to 28 days before dosing), dosing on Day 1, a post-dose period (Days 5 to 57) and a final follow-up visit on Day 71. A total of 54 participants were enrolled in the study.
Groups:
- Cohort 1: VIS954 Dose 1: Participants received a single dose of VIS954 at Dose 1 via subcutaneous (SC) injection on Day 1.
- Cohort 2: VIS954 Dose 2: Participants received a single dose of VIS954 at Dose 2 via SC injection on Day 1.
- Cohort 3: VIS954 Dose 3: Participants received a single dose of VIS954 at Dose 3 via SC injection on Day 1.
- Cohort 4: VIS954 Dose 4: Participants received a single dose of VIS954 at Dose 4 via SC injection on Day 1.
- Cohort 5: VIS954 Dose 5: Participants received a single dose of VIS954 at Dose 5 via SC injection on Day 1.
- Cohort 6: VIS954 Dose 6: Participants received a single dose of VIS954 at Dose 6 via SC injection on Day 1.
- Cohort 1 to 6: Pooled Placebo: Participants received a single dose of placebo matched to VIS954 via SC injection on Day 1.
Period: Overall Study
Arm/Group | Cohort 1: VIS954 Dose 1 | Cohort 2: VIS954 Dose 2 | Cohort 3: VIS954 Dose 3 | Cohort 4: VIS954 Dose 4 | Cohort 5: VIS954 Dose 5 | Cohort 6: VIS954 Dose 6 | Cohort 1 to 6: Pooled Placebo
Started | 7 | 7 | 7 | 7 | 7 | 7 | 12
Completed | 7 | 7 | 7 | 7 | 7 | 7 | 12
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all participants who received trial intervention (active or placebo).
Groups:
- Cohort 1: VIS954 Dose 1: Participants received a single dose of VIS954 at Dose 1 via SC injection on Day 1.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: VIS954 Dose 1 | Cohort 2: VIS954 Dose 2 | Cohort 3: VIS954 Dose 3 | Cohort 4: VIS954 Dose 4 | Cohort 5: VIS954 Dose 5 | Cohort 6: VIS954 Dose 6 | Cohort 1 to 6: Pooled Placebo | Total
Number analyzed (Participants) | 7 | 7 | 7 | 7 | 7 | 7 | 12 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.4 (8.2) | 40.6 (8.1) | 38.9 (9.6) | 39.0 (7.7) | 39.4 (9.3) | 39.0 (10.2) | 36.5 (7.6) | 38.2 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 4 | 4 | 2 | 3 | 7 | 29
  Male | 2 | 3 | 3 | 3 | 5 | 4 | 5 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 2 | 1 | 2 | 3 | 10
  Not Hispanic or Latino | 6 | 6 | 7 | 5 | 6 | 5 | 9 | 44
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 1 | 3 | 2 | 1 | 0 | 0 | 4 | 11
  Asian | 4 | 3 | 2 | 4 | 6 | 3 | 1 | 23
  White | 2 | 1 | 1 | 1 | 1 | 3 | 5 | 14
  Other | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
  Multiple | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. A serious adverse event (SAE) was any untoward medical occurrence that, at any dose, resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, was a suspected transmission of any infectious agent via an authorized medicinal product or was an important medical event that jeopardized the participant or required medical or surgical intervention to prevent 1 of the other outcomes listed above. TEAEs were AEs that first occurred or worsened in severity after the study intervention administration, and up to Day 71 (including the follow-up period) after the study intervention administration.
Time Frame: From study intervention administration (Day 1) up to end of follow-up (Day 71)
Population: The safety analysis set included all participants who received trial intervention (active or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: VIS954 Dose 1 | Cohort 2: VIS954 Dose 2 | Cohort 3: VIS954 Dose 3 | Cohort 4: VIS954 Dose 4 | Cohort 5: VIS954 Dose 5 | Cohort 6: VIS954 Dose 6 | Cohort 1 to 6: Pooled Placebo
Number analyzed (Participants) | 7 | 7 | 7 | 7 | 7 | 7 | 12
Participants
  TEAEs | 2 | 1 | 1 | 1 | 3 | 2 | 4
  TESAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Wong-Baker FACES Pain Rating Scale
Description: The Wong-Baker FACES Pain Rating Scale was a subjective self-report that was used to record each participant's perception of pain associated with their injection. The scale ranged from 0 to 10 and showed a series of faces ranging from a happy face at 0 which represented "no hurt" to a crying face at 10 which represented "hurts worst." Based on the faces and descriptions, the participant recorded their level of pain. Higher scores indicated more severe pain.
Time Frame: Day 1 (1 and 4 hours post-dose), Day 2 (24 hours post-dose), and on Days 3 and 29
Population: The safety analysis set included all participants who received trial intervention (active or placebo).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cohort 1: VIS954 Dose 1 | Cohort 2: VIS954 Dose 2 | Cohort 3: VIS954 Dose 3 | Cohort 4: VIS954 Dose 4 | Cohort 5: VIS954 Dose 5 | Cohort 6: VIS954 Dose 6 | Cohort 1 to 6: Pooled Placebo
Number analyzed (Participants) | 7 | 7 | 7 | 7 | 7 | 7 | 12
units on a scale
  Day 1: 1 hour post-dose | 0 (0) | 0 (0) | 0 (0) | 0.3 (0.8) | 0 (0) | 0 (0) | 0.3 (1.2)
  Day 1: 4 hours post-dose | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0.3 (1.2)
  Day 2: 24 hours post-dose | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Day 3 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Day 29 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

3. Secondary Outcome: Maximum Serum Concentration (Cmax) of VIS954
Description: Blood samples were collected for measurement of serum concentrations of VIS954 at the specified time points from Day 1 (within 2 hours pre-dose) to Day 71. The pharmacokinetic (PK) parameters of VIS954 were derived using noncompartmental analysis method.
Time Frame: Day 1 (within 2 hours pre-dose) and at multiple timepoints post-dose up to Day 71
Population: PK analysis set: participants who received VIS954 and had at least 1 measured post-dose VIS954 serum concentration at scheduled PK time after start of dosing for at least 1 PK analyte without protocol deviations/events with potential to affect evaluation of PK data. As pre-specified in SAP, 13 participants (7 and 6 in Cohorts 1 and 2) were excluded from PK analysis as PK profiles were below limit of quantitation (BLQ). Only participants with data collected at specified timepoints are reported.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (mcg/mL)
Arm/Group | Cohort 1: VIS954 Dose 1 | Cohort 2: VIS954 Dose 2 | Cohort 3: VIS954 Dose 3 | Cohort 4: VIS954 Dose 4 | Cohort 5: VIS954 Dose 5 | Cohort 6: VIS954 Dose 6
Number analyzed (Participants) | 0 | 1 | 7 | 6 | 7 | 7
micrograms per milliliter (mcg/mL) |  | 0.0660 (NA) — NA indicates that the standard deviation (SD) was not estimable for 1 participant. | 1.961 (1.378) | 4.423 (2.851) | 16.82 (12.95) | 32.61 (12.00)

4. Secondary Outcome: Time of Maximum Serum Concentration (Tmax) of VIS954
Description: Blood samples were collected for measurement of serum concentrations of VIS954 at the specified time points from Day 1 (within 2 hours pre-dose) to Day 71. The PK parameters of VIS954 were derived using noncompartmental analysis method.
Time Frame: Day 1 (within 2 hours pre-dose) and at multiple timepoints post-dose up to Day 71
Population: The PK analysis set included all participants who received VIS954 and had at least 1 measured post-dose VIS954 serum concentration at scheduled PK time after start of dosing for at least 1 PK analyte without protocol deviations or events with potential to affect the evaluation of the PK data. As pre-specified in SAP, 13 participants (7 and 6 in Cohorts 1 and 2) were excluded from PK analysis as PK profiles were BLQ. Only participants with data collected at specified timepoints are reported.
Measure: Median (Full Range); unit: hour
Arm/Group | Cohort 1: VIS954 Dose 1 | Cohort 2: VIS954 Dose 2 | Cohort 3: VIS954 Dose 3 | Cohort 4: VIS954 Dose 4 | Cohort 5: VIS954 Dose 5 | Cohort 6: VIS954 Dose 6
Number analyzed (Participants) | 0 | 1 | 7 | 6 | 7 | 7
hour |  | 48.00 [48.00 to 48.00] | 48.00 [4.02 to 98.35] | 71.82 [48.00 to 166.38] | 74.02 [72.12 to 169.70] | 95.60 [48.00 to 169.70]

5. Secondary Outcome: Area Under the Concentration-Time Curve From Pre-dose Extrapolated to Infinite Time (AUC0-inf) of VIS954
Description: as for outcome 4
Time Frame: Day 1 (within 2 hours pre-dose) and at multiple timepoints post-dose up to Day 71
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: hour*mcg/mL
Arm/Group | Cohort 1: VIS954 Dose 1 | Cohort 2: VIS954 Dose 2 | Cohort 3: VIS954 Dose 3 | Cohort 4: VIS954 Dose 4 | Cohort 5: VIS954 Dose 5 | Cohort 6: VIS954 Dose 6
Number analyzed (Participants) | 0 | 0 | 1 | 3 | 4 | 7
hour*mcg/mL |  |  | 395 (NA) — NA indicates that the SD was not estimable for 1 participant. | 1463 (1324) | 5529 (1877) | 11560 (5503)

6. Secondary Outcome: Area Under the Concentration-Time Curve From Pre-dose to the Last Quantifiable Concentration (AUC0-last) of VIS954
Description: as for outcome 4
Time Frame: Day 1 (within 2 hours pre-dose) and at multiple timepoints post-dose up to Day 71
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: hour*mcg/mL
Arm/Group | Cohort 1: VIS954 Dose 1 | Cohort 2: VIS954 Dose 2 | Cohort 3: VIS954 Dose 3 | Cohort 4: VIS954 Dose 4 | Cohort 5: VIS954 Dose 5 | Cohort 6: VIS954 Dose 6
Number analyzed (Participants) | 0 | 1 | 7 | 6 | 7 | 7
hour*mcg/mL |  | 3.17 (NA) — NA indicates that the SD was not estimable for 1 participant. | 188.4 (151.2) | 872.4 (974.1) | 3604 (2684) | 11470 (5458)

7. Secondary Outcome: Apparent Terminal Elimination Half-Life (t1/2) of VIS954
Description: as for outcome 4
Time Frame: Day 1 (within 2 hours pre-dose) and at multiple timepoints post-dose up to Day 71
Population: as for outcome 4
Measure: Median (Full Range); unit: hour
Arm/Group | Cohort 1: VIS954 Dose 1 | Cohort 2: VIS954 Dose 2 | Cohort 3: VIS954 Dose 3 | Cohort 4: VIS954 Dose 4 | Cohort 5: VIS954 Dose 5 | Cohort 6: VIS954 Dose 6
Number analyzed (Participants) | 0 | 0 | 2 | 3 | 4 | 7
hour |  |  | 85.25 [37.5 to 133] | 33.6 [25.8 to 105] | 48.0 [41.3 to 82.4] | 76.3 [44.7 to 101]

8. Secondary Outcome: Apparent Volume of Distribution (Vd/F) of VIS954
Description: as for outcome 4
Time Frame: Day 1 (within 2 hours pre-dose) and at multiple timepoints post-dose up to Day 71
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: liter
Arm/Group | Cohort 1: VIS954 Dose 1 | Cohort 2: VIS954 Dose 2 | Cohort 3: VIS954 Dose 3 | Cohort 4: VIS954 Dose 4 | Cohort 5: VIS954 Dose 5 | Cohort 6: VIS954 Dose 6
Number analyzed (Participants) | 0 | 0 | 1 | 3 | 4 | 7
liter |  |  | 12.3 (NA) — NA indicates that the SD was not estimable for 1 participant. | 10.12 (1.797) | 5.218 (1.606) | 8.536 (5.579)

9. Secondary Outcome: Apparent Clearance After Extravascular Dosing (CL/F) of VIS954
Description: as for outcome 4
Time Frame: Day 1 (within 2 hours pre-dose) and at multiple timepoints post-dose up to Day 71
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: liter per hour
Arm/Group | Cohort 1: VIS954 Dose 1 | Cohort 2: VIS954 Dose 2 | Cohort 3: VIS954 Dose 3 | Cohort 4: VIS954 Dose 4 | Cohort 5: VIS954 Dose 5 | Cohort 6: VIS954 Dose 6
Number analyzed (Participants) | 0 | 0 | 1 | 3 | 4 | 7
liter per hour |  |  | 0.228 (NA) — NA indicates that the SD was not estimable for 1 participant. | 0.1864 (0.1108) | 0.06911 (0.02358) | 0.07976 (0.05542)

10. Secondary Outcome: Time Spent Above 40 Percentage Receptor Occupancy (RO) for Neutrophils
Description: Blood samples were collected at the specified time points to characterize the effect of VIS954 binding. The time spent above 40% RO was defined as duration in hours from date and time of dosing until the date and time of pharmacodynamic (PD) collection when %RO >40%. Baseline was defined as the last non-missing measurement taken prior to reference start date (including unscheduled assessments).
Time Frame: Baseline (Day -1) up to Day 71
Population: The PD analysis set included all participants who received trial intervention (active or placebo) and had at least 1 measured PD value at a scheduled time point after start of dosing.
Measure: Median (Full Range); unit: hour
Arm/Group | Cohort 1: VIS954 Dose 1 | Cohort 2: VIS954 Dose 2 | Cohort 3: VIS954 Dose 3 | Cohort 4: VIS954 Dose 4 | Cohort 5: VIS954 Dose 5 | Cohort 6: VIS954 Dose 6 | Cohort 1 to 6: Pooled Placebo
Number analyzed (Participants) | 7 | 7 | 7 | 7 | 7 | 7 | 12
hour | 0.0 [0.0 to 0.0] | 48.0 [0.0 to 74.1] | 239.2 [215.8 to 314.1] | 335.5 [239.7 to 671.4] | 503.1 [217.0 to 673.7] | 1008.1 [838.9 to 1680.0] | 0.0 [0.0 to 0.0]

ADVERSE EVENTS:
Time Frame: From study intervention administration (Day 1) up to end of follow-up (Day 71)
Description: The safety analysis set included all participants who received trial intervention (active or placebo).
Arm/Group | Cohort 1: VIS954 Dose 1 | Cohort 2: VIS954 Dose 2 | Cohort 3: VIS954 Dose 3 | Cohort 4: VIS954 Dose 4 | Cohort 5: VIS954 Dose 5 | Cohort 6: VIS954 Dose 6 | Cohort 1 to 6: Pooled Placebo
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7 | 0/7 | 0/7 | 0/7 | 0/7 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7 | 0/7 | 0/7 | 0/7 | 0/7 | 0/12
Other Adverse Events (participants affected / at risk) | 2/7 | 1/7 | 1/7 | 1/7 | 3/7 | 2/7 | 4/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: VIS954 Dose 1 (N=7) | Cohort 2: VIS954 Dose 2 (N=7) | Cohort 3: VIS954 Dose 3 (N=7) | Cohort 4: VIS954 Dose 4 (N=7) | Cohort 5: VIS954 Dose 5 (N=7) | Cohort 6: VIS954 Dose 6 (N=7) | Cohort 1 to 6: Pooled Placebo (N=12)
Blood loss anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Injection site bruising (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injection site pruritus (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Injection site reaction (General disorders) | 0 | 0 | 0 | 1 | 2 | 1 | 3
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-10-20): https://cdn.clinicaltrials.gov/large-docs/04/NCT06212804/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-23): https://cdn.clinicaltrials.gov/large-docs/04/NCT06212804/SAP_001.pdf